CLINICAL TRIAL: NCT06981273
Title: SPAIN Trial Comparing Open vs Robotic Pancreatoduodenectomy
Brief Title: Robotic vs Open Pancreatoduodenectomy
Acronym: SPAIN PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Benedetto Ielpo, prof, Hospital del Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPAIN PD Trial
Record Dates: First submitted 2025-03-16; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Pancreas Neoplasms
Keywords: Robotic; pancreaticoduodenectony; Robotic surgery
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic (Experimental): Robotic pancreatoduodenectomy is performed under the robotic da Vinci system where at least the pancreatic and biliary anastomosis is performed throughout this approach.
  Interventions: Procedure: Robotic pancreatoduodenectomy
- Open (Active Comparator): open pancreatoduodenectomy is performed through a laparotomy following the standard criteria for this type of surgery.
  Interventions: Procedure: open pancreatoduodenectomy

INTERVENTIONS:
Procedure: Robotic pancreatoduodenectomy — A Robotic approach pancreatoduodenectomy is performed on patients
  Arms: Robotic
Procedure: open pancreatoduodenectomy — An open approach for pancreatoduodenectomy is performed
  Arms: Open

SUMMARY:
Pancreatic surgery, specifically pancreatoduodenectomy (PD), is a complex procedure often required for patients with pancreatic or other periampullary cancers. In recent years, minimally invasive techniques have become more popular, especially robotic-assisted surgery. However, there are limited studies comparing robotic surgery to traditional open surgery.

This is a national, multicenter study in Spain comparing the outcomes of robotic versus open pancreatoduodenectomy (PD). The main goal is to assess complications within 90 days after surgery. This study is important because it will provide evidence on which approach is safer and more effective for patients.

The study follows a **prospective, randomized, and multicenter design**, meaning patients are assigned to either robotic or open surgery randomly, and multiple hospitals are involved. The study will include all eligible patients undergoing planned PD surgery, either by robotic or open technique.

To be included in the study, patients must meet these conditions:

* Be **18 years or older**.
* Require **planned PD surgery**.
* Sign an **informed consent form**.

Who Cannot Participate?

Patients will **not** be included if they:

* **Refuse the procedure**.
* Have **uncertainty about vascular involvement**.
* Have a severe health condition classified as **ASA IV** (high-risk for surgery).

The main outcome measured will be the **Comprehensive Complication Index (CCI), a standardized way to assess post-surgical complications. Additional factors being studied include:

* **Clinical outcomes** during and after surgery.
* **Quality of life** assessments.
* **Surgical costs**.
* **Hospital stay duration**.
* **Need to switch from robotic to open surgery**.
* **Need for additional surgery (reoperations)**.
* **Hospital readmissions**.

Where Is the Study Being Conducted?

The study is being conducted in **ten major hospitals across Spain**:

1. Hospital del Mar, Barcelona
2. Hospital Balmis, Alicante
3. Hospital Vall d'Hebron, Barcelona
4. Arnau de Vilanova, Lleida
5. Joan XXIII, Tarragona
6. Hospital Sant Pau, Barcelona
7. Germans Trias i Pujol, Barcelona
8. Hospital Clínic, Barcelona
9. HM Sanchinarro, Madrid
10. Hospital Rio Hortega, Valladolid

How Long Will the Study Last? The study will take **two years** to complete, and patients will be followed for **three years** after surgery to track long-term outcomes.

Why Is This Study Important for Patients? For patients undergoing PD, this study will provide essential information about the risks and benefits of robotic versus open surgery. The findings will help doctors determine the best surgical approach, leading to improved safety, faster recovery, and better long-term health outcomes.

If you are a patient facing this type of surgery, participating in this study could contribute to valuable medical knowledge while ensuring that you receive a carefully monitored treatment plan.

DETAILED DESCRIPTION:
Introduction

Pancreatoduodenectomy (PD), commonly known as the Whipple procedure, is a complex surgical procedure used to treat pancreatic, bile duct, and duodenal diseases, including cancer. Traditionally, this surgery has been performed using an open approach (PDA), but recent advancements in minimally invasive techniques have introduced the robotic approach (PDR) as a potential alternative.

Minimally invasive robotic surgery may offer benefits such as reduced blood loss, shorter hospital stays, and potentially lower complication rates. However, there is limited high-quality evidence comparing the outcomes of robotic PD versus open PD. This national, multicenter, randomized clinical trial aims to provide clear answers by analyzing postoperative complications and overall patient outcomes.

Primary Objective

Evaluate postoperative complications using the CCI within 90 days after surgery.

Objectives This clinical trial aims to compare two different surgical approaches, PDR and PDA, in relation to postoperative morbidity within 90 days following surgery. Morbidity is assessed using the Complication Index (CCI) (www.assesssurgery.com). The primary objective is to measure CCI®, which tracks complications up to 90 days after surgery. Secondary objectives include intraoperative variables (e.g., blood loss, operative time, and conversion), postoperative morbidity (e.g., pancreatic-specific complications as defined by ISGPS), oncological outcomes in cases of malignancy (radicality, lymph node removal, and time until adjuvant chemotherapy), healthcare resource utilization (length of stay, readmissions, ICU stay), and quality of life and recovery post-surgery.

Secondary Objectives

Intraoperative outcomes: Blood loss, operative time, and conversion rates from robotic to open surgery.

Postoperative morbidity: Evaluated using the International Study Group of Pancreatic Surgery (ISGPS) definitions.

Oncological outcomes (for cancer patients): Tumor clearance, number of lymph nodes removed, and time to adjuvant chemotherapy.

Healthcare resource utilization: Hospital stay, ICU admission, and hospital readmissions.

Quality of life and recovery after surgery.

Hypothesis The PDR surgical procedure demonstrates non-inferiority in the post-operative CCI score up to 90 days after surgery.

Materials and Methods

Study Design

This is a national, multicenter, randomized, prospective clinical trial with parallel groups comparing patients undergoing PD for any cause. Patients will be randomized into two groups:

Group 1: PDR Group 2: PDA The study will span 2 years. The research will be conducted in centers with an annual volume of at least 30 pancreatic resections (distal and cephalic) and surgeons with personal experience of at least 20 PDRs annually. A minimum of 30 pancreatic resections includes at least 20 pancreatoduodenectomies annually.

Sample Size This is a non-inferiority study. According to previous studies, a clinically relevant mean difference in CCI is 7.5, while the average standard deviation is approximately 20 in major abdominal surgeries. A total of 93 patients will need to be enrolled in the trial (46 and 47 per group), accounting for a 5% dropout rate, with an alpha error of 5% and a beta error of 20%.

Data Collection

Clinical Data Postoperative complications will be classified and evaluated according to the Clavien-Dindo classification (I to V) and the CCI numeric scale (www.assesssurgery.com). Major complications are those rated IIIa or higher. Complications, readmissions, and mortality will be measured up to 90 days.

Safety Assessment of Procedures

Both techniques, PDR and PDA, will be evaluated for adverse events. The following complications will be recorded in the Clinical Data Record (CRD):

Blood loss and need for transfusion during the procedure Postoperative hemorrhage Postoperative transfusion Biliary fistula Need for re-intervention Need for readmission Postoperative death Economic Data Economic data will be collected based on the single cost assigned to each procedure, calculated using the RECH system (Spanish Hospital Cost Network: https://www.rechosp.org). The costs will be derived from the National Health System's (SNS) diagnostic-related groups (DRG). The total cost will be calculated by multiplying the number of resource units used by the unit cost.

Measures to Minimize Bias Two main limitations are anticipated. The first concerns variability in surgical techniques among the surgeons. To minimize this, a meeting of all participating centers will be held to standardize surgical techniques. Furthermore, quality control will involve sending a video of the PDR procedure from each surgeon for evaluation.

The second limitation relates to patient recruitment. To address this, a conservative estimate of potential candidates was made, and centers with high volumes of pancreatic resections (at least 30 per year, including 20 pancreatoduodenectomies) have been selected.

Randomization Randomization will be performed using block assignment stratified by center, ensuring balanced groups within each participating hospital. Randomization between the robotic and open arms will occur before surgery with a 1:1 ratio using an online system.

Blinding This study will be single-blinded, meaning patients will not be aware of which group they belong to. After surgery, a cover will be applied to the abdominal wall so patients cannot see whether they had a robotic or open procedure.

Surgical Procedures

PDA:

The procedure begins with a bilateral subcostal incision. After initial exploration, if no distant disease is found, a PD will be performed. Reconstruction follows after the surgical specimen is removed.

PDR:

The procedure starts with robotic trocar placement, along with up to two additional laparoscopic trocars. Surgical steps follow the PDA procedure, but the specimen is removed through a mini-incision. Hybrid techniques (laparoscopic resection and robotic reconstruction) are excluded.

Data Recording Study variables will be stored in an online data collection form (CRD), which will automatically transfer data to a database. The system used for this will be Red Cap. The investigators and study monitor will have digital access to the Red Cap database to include new patients and review data during follow-up. Patient names will not appear in the database to ensure confidentiality. A subject code will be used for anonymity, and an identification register will link the code to the patient's medical record.

Statistical Analysis Data will be analyzed using IBM SPSS Statistics for Windows version 24.0 (IBM Corp.). Statistical tests such as Student's T-test, Mann-Whitney U test, Chi-square, and Fisher's exact test will be employed. Categorical data will be presented as frequency and percentage, and continuous data as mean, standard deviation, or median with interquartile range. Subgroups will be analyzed using Chi-square, Mann-Whitney U, and Kruskal-Wallis tests, with p<0.05 indicating statistical significance.

Ethical Aspects The study will be registered on www.controlled-trials.com and will follow the ethical principles of the Declaration of Helsinki (2013) and Good Clinical Practice (GCP). Informed consent will be obtained from all participants, and the study will be reviewed by an Ethics Committee. The protocol will be registered on clinicaltrial.gov. Confidentiality will be maintained, and data will not be shared with third parties without consent.

Sample Management and Confidentiality Only necessary biological samples will be taken, with all patient data stored pseudonymized to ensure confidentiality. The study will comply with GDPR and local privacy laws.

Funding Funding for the study will be requested from the Spanish Association of Surgeons (AEC) for a total of €10,000, which will be used for insurance and monitoring.

Monitoring and Auditing The study will be monitored by clinical investigators and a data manager for periodic center audits.

Public Disclosure and Publication Results will be submitted to a high-impact medical journal, with authorship based on participant center recruitment volume. The study's findings will also be published in scientific journals following local regulations.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Patients requiring planned pancreatoduodenectomy (robotic or open).
* Signed informed consent to participate in the study.

Exclusion Criteria:

* Patients who refuse the procedure.
* Uncertainty about vascular involvement that could affect resectability.
* Poor general health status (American Society of Anesthesiologists [ASA] classification IV).
* Pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Complication Index | up to 90 days after surgery
  Morbidity is assessed using the Complication Index (CCI) (www.assesssurgery.com). The primary objective is to measure CCI®, which tracks complications up to 90 days after surgery.

SECONDARY OUTCOMES:
Cost effectiveness | 3 months after surgery
  Economic data will be collected based on the single cost assigned to each procedure, calculated using the RECH system (Spanish Hospital Cost Network: https://www.rechosp.org). The costs will be derived from the National Health System's (SNS) diagnostic-related groups (DRG). The total cost will be calculated by multiplying the number of resource units used by the unit cost.
  Effectiveness will be used with the EQ-5D-5L using the QALY model
Tumor clearance | until the end of the study
  pancreatic stump margins defined as R0, R1 or R2
operative time | during the surgery
  Duration of the operation in minutes.
Blood loss | during the surgery
  intraoperative blood loss in ml
Conversion to open surgery | during surgery
  This is only for the robotic approach where conversion to open occurred
Pancreatic Fistula | after surgery up to 90 days from operation
  collection of data of pancreatic fistula according to International Study Group of Pancreatic Surgery (ISGPS) : Type A, B or C
EORTC QLQ-C30 | before and after surgery at 30 and 90 days
  scale of quality if life
QoR-15 | after surgery at 30 and 90 days
  test of quality of recuperation after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
I do not want to be contacted by commercial industry regarding this study

REFERENCES:
- [Background] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Background] Slankamenac K, Nederlof N, Pessaux P, de Jonge J, Wijnhoven BP, Breitenstein S, Oberkofler CE, Graf R, Puhan MA, Clavien PA. The comprehensive complication index: a novel and more sensitive endpoint for assessing outcome and reducing sample size in randomized controlled trials. Ann Surg. 2014 Nov;260(5):757-62; discussion 762-3. doi: 10.1097/SLA.0000000000000948. PMID 25379846
- [Background] van Hilst J, de Graaf N, Abu Hilal M, Besselink MG. The Landmark Series: Minimally Invasive Pancreatic Resection. Ann Surg Oncol. 2021 Mar;28(3):1447-1456. doi: 10.1245/s10434-020-09335-3. Epub 2020 Dec 19. PMID 33341916
- [Background] Boggi U, Signori S, De Lio N, Perrone VG, Vistoli F, Belluomini M, Cappelli C, Amorese G, Mosca F. Feasibility of robotic pancreaticoduodenectomy. Br J Surg. 2013 Jun;100(7):917-25. doi: 10.1002/bjs.9135. PMID 23640668
- [Background] Tran TB, Dua MM, Worhunsky DJ, Poultsides GA, Norton JA, Visser BC. The First Decade of Laparoscopic Pancreaticoduodenectomy in the United States: Costs and Outcomes Using the Nationwide Inpatient Sample. Surg Endosc. 2016 May;30(5):1778-83. doi: 10.1007/s00464-015-4444-y. Epub 2015 Aug 15. PMID 26275542
- [Background] Jones LR, Zwart MJW, Molenaar IQ, Koerkamp BG, Hogg ME, Hilal MA, Besselink MG. Robotic Pancreatoduodenectomy: Patient Selection, Volume Criteria, and Training Programs. Scand J Surg. 2020 Mar;109(1):29-33. doi: 10.1177/1457496920911815. PMID 32192422
- [Background] van Hilst J, de Rooij T, Bosscha K, Brinkman DJ, van Dieren S, Dijkgraaf MG, Gerhards MF, de Hingh IH, Karsten TM, Lips DJ, Luyer MD, Busch OR, Festen S, Besselink MG; Dutch Pancreatic Cancer Group. Laparoscopic versus open pancreatoduodenectomy for pancreatic or periampullary tumours (LEOPARD-2): a multicentre, patient-blinded, randomised controlled phase 2/3 trial. Lancet Gastroenterol Hepatol. 2019 Mar;4(3):199-207. doi: 10.1016/S2468-1253(19)30004-4. Epub 2019 Jan 24. PMID 30685489
- [Background] Wang M, Li D, Chen R, Huang X, Li J, Liu Y, Liu J, Cheng W, Chen X, Zhao W, Li J, Tan Z, Huang H, Li D, Zhu F, Qin T, Ma J, Yu G, Zhou B, Zheng S, Tang Y, Han W, Meng L, Ke J, Feng F, Chen B, Yin X, Chen W, Ma H, Xu J, Liu Y, Lin R, Dong Y, Yu Y, Liu J, Zhang H, Qin R; Minimally Invasive Treatment Group in the Pancreatic Disease Branch of China's International Exchange and Promotion Association for Medicine and Healthcare (MITG-P-CPAM). Laparoscopic versus open pancreatoduodenectomy for pancreatic or periampullary tumours: a multicentre, open-label, randomised controlled trial. Lancet Gastroenterol Hepatol. 2021 Jun;6(6):438-447. doi: 10.1016/S2468-1253(21)00054-6. Epub 2021 Apr 27. PMID 33915091
- [Background] Poves I, Burdio F, Morato O, Iglesias M, Radosevic A, Ilzarbe L, Visa L, Grande L. Comparison of Perioperative Outcomes Between Laparoscopic and Open Approach for Pancreatoduodenectomy: The PADULAP Randomized Controlled Trial. Ann Surg. 2018 Nov;268(5):731-739. doi: 10.1097/SLA.0000000000002893. PMID 30138162
- [Background] Kendrick ML, van Hilst J, Boggi U, de Rooij T, Walsh RM, Zeh HJ, Hughes SJ, Nakamura Y, Vollmer CM, Kooby DA, Asbun HJ; Minimally Invasive Pancreatic Resection Organizing Committee. Minimally invasive pancreatoduodenectomy. HPB (Oxford). 2017 Mar;19(3):215-224. doi: 10.1016/j.hpb.2017.01.023. PMID 28317658
- [Background] de Rooij T, van Hilst J, Topal B, Bosscha K, Brinkman DJ, Gerhards MF, de Hingh IH, Karsten TM, Lips DJ, Luyer MD, Marsman HA, van Rijssen LB, Steen MW, Busch OR, Festen S, Besselink MG; Dutch Pancreatic Cancer Group. Outcomes of a Multicenter Training Program in Laparoscopic Pancreatoduodenectomy (LAELAPS-2). Ann Surg. 2019 Feb;269(2):344-350. doi: 10.1097/SLA.0000000000002563. PMID 29099400
- [Background] de Rooij T, Lu MZ, Steen MW, Gerhards MF, Dijkgraaf MG, Busch OR, Lips DJ, Festen S, Besselink MG; Dutch Pancreatic Cancer Group. Minimally Invasive Versus Open Pancreatoduodenectomy: Systematic Review and Meta-analysis of Comparative Cohort and Registry Studies. Ann Surg. 2016 Aug;264(2):257-67. doi: 10.1097/SLA.0000000000001660. PMID 26863398
- [Background] Jin T, Altaf K, Xiong JJ, Huang W, Javed MA, Mai G, Liu XB, Hu WM, Xia Q. A systematic review and meta-analysis of studies comparing laparoscopic and open distal pancreatectomy. HPB (Oxford). 2012 Nov;14(11):711-24. doi: 10.1111/j.1477-2574.2012.00531.x. Epub 2012 Aug 7. PMID 23043660
- [Background] Klotz R, Mihaljevic AL, Kulu Y, Sander A, Klose C, Behnisch R, Joos MC, Kalkum E, Nickel F, Knebel P, Pianka F, Diener MK, Buchler MW, Hackert T. Robotic versus open partial pancreatoduodenectomy (EUROPA): a randomised controlled stage 2b trial. Lancet Reg Health Eur. 2024 Feb 22;39:100864. doi: 10.1016/j.lanepe.2024.100864. eCollection 2024 Apr. PMID 38420108
- [Background] de Graaf N, Emmen AMLH, Ramera M, Bjornsson B, Boggi U, Bruna CL, Busch OR, Daams F, Ferrari G, Festen S, van Hilst J, D'Hondt M, Ielpo B, Keck T, Khatkov IE, Koerkamp BG, Lips DJ, Luyer MDP, Mieog JSD, Morelli L, Molenaar IQ, van Santvoort HC, Sprangers MAG, Ferrari C, Berkhof J, Maisonneuve P, Abu Hilal M, Besselink MG; European Consortium on Minimally Invasive Pancreatic Surgery (E-MIPS). Minimally invasive versus open pancreatoduodenectomy for pancreatic and peri-ampullary neoplasm (DIPLOMA-2): study protocol for an international multicenter patient-blinded randomized controlled trial. Trials. 2023 Oct 12;24(1):665. doi: 10.1186/s13063-023-07657-7. PMID 37828593
- [Background] Asbun HJ, Moekotte AL, Vissers FL, Kunzler F, Cipriani F, Alseidi A, D'Angelica MI, Balduzzi A, Bassi C, Bjornsson B, Boggi U, Callery MP, Del Chiaro M, Coimbra FJ, Conrad C, Cook A, Coppola A, Dervenis C, Dokmak S, Edil BH, Edwin B, Giulianotti PC, Han HS, Hansen PD, van der Heijde N, van Hilst J, Hester CA, Hogg ME, Jarufe N, Jeyarajah DR, Keck T, Kim SC, Khatkov IE, Kokudo N, Kooby DA, Korrel M, de Leon FJ, Lluis N, Lof S, Machado MA, Demartines N, Martinie JB, Merchant NB, Molenaar IQ, Moravek C, Mou YP, Nakamura M, Nealon WH, Palanivelu C, Pessaux P, Pitt HA, Polanco PM, Primrose JN, Rawashdeh A, Sanford DE, Senthilnathan P, Shrikhande SV, Stauffer JA, Takaori K, Talamonti MS, Tang CN, Vollmer CM, Wakabayashi G, Walsh RM, Wang SE, Zinner MJ, Wolfgang CL, Zureikat AH, Zwart MJ, Conlon KC, Kendrick ML, Zeh HJ, Hilal MA, Besselink MG; International Study Group on Minimally Invasive Pancreas Surgery (I-MIPS). The Miami International Evidence-based Guidelines on Minimally Invasive Pancreas Resection. Ann Surg. 2020 Jan;271(1):1-14. doi: 10.1097/SLA.0000000000003590. PMID 31567509
- [Background] Wente MN, Veit JA, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Yeo CJ, Buchler MW. Postpancreatectomy hemorrhage (PPH): an International Study Group of Pancreatic Surgery (ISGPS) definition. Surgery. 2007 Jul;142(1):20-5. doi: 10.1016/j.surg.2007.02.001. PMID 17629996
- [Background] Hirata K, Egawa S, Kimura Y, Nobuoka T, Oshima H, Katsuramaki T, Mizuguchi T, Furuhata T. Current status of surgery for pancreatic cancer. Dig Surg. 2007;24(2):137-47. doi: 10.1159/000102067. Epub 2007 Apr 27. PMID 17476103
- [Background] Matsuno S, Egawa S, Fukuyama S, Motoi F, Sunamura M, Isaji S, Imaizumi T, Okada S, Kato H, Suda K, Nakao A, Hiraoka T, Hosotani R, Takeda K. Pancreatic Cancer Registry in Japan: 20 years of experience. Pancreas. 2004 Apr;28(3):219-30. doi: 10.1097/00006676-200404000-00002. PMID 15084961